CLINICAL TRIAL: NCT02351583
Title: Microcirculatory and Tissue and Cerebral Oxygenation Differences Between Preeclampsia and Normal Pregnancy: An Observation Study
Brief Title: Microcirculatory and Tissue and Cerebral Oxygenation in Preeclampsia and Normal Pregnancy: An Observation Study
Status: Withdrawn | Type: Observational
Why Stopped: equipment difficulties
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mohamed Tiouririne, MD, Associate Professor, Anesthesiology, University of Virginia
Other Study IDs: 17837
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy; Eclampsia
MeSH Terms: conditions — Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- preclampsia: 10 with diagnosis of preeclampsia will be examined with both NIRS and cytocam to obtain data
  Interventions: Device: CytoCam; Device: NIRS Artinis PortaLite with OxySoft softwear
- normal pregnancy: 10 with normal pregnancy will be examined with both NIRS and cytocam to obtain data
  Interventions: Device: CytoCam; Device: NIRS Artinis PortaLite with OxySoft softwear

INTERVENTIONS:
Device: CytoCam — The side-stream darkfield camera ( CytoCam) will be put under the subjects tongue for 5-10 minutes. Multiple pictures of the small blood vessels will be taken.
Device: NIRS Artinis PortaLite with OxySoft softwear — . The NIRS probe will be applied to one of the patient's thenar muscle and over the patient forehead and tissue oxygenation (TOI) will be recorded for 5 minutes.

SUMMARY:
Preeclampsia is a disease of pregnancy affecting 3% to 8% of all pregnancies and is a major cause of maternal and perinatal morbidity and mortality. Characterized by alter placentation with subsequent release of inflammatory mediators leading to a generalized endothelial dysfunction. It is now accepted that endothelial dysfunction heralds the clinical manifestations of preeclampsia.

The side-stream darkfield (SDF) microscopy device emits a 550 nm green light with a depth region of interest of 500 um. Green light is absorbed by the erythrocytes and appears black. SDF is a well-known non-invasive tool that can study the microcirculatory changes. It was used before in many situations especially in sepsis and septic shock patients.

Near-infra-red spectroscopy (NIRS) device, measures the absorbance of near-infra-red (NIR) light by tissues perfused with oxygenated blood, and is capable of measuring changes in parenchymal volume tissues. It was used before in many situations (including pregnant patients) to reflect the tissue oxygenations.

The investigators are planning to use the SDF and NIRS tools to study the microcirculatory change in preeclamptic subjects and normal pregnant subjects. If these two devices are able to determine any changes this should stand as a baseline for future studies in this field.

DETAILED DESCRIPTION:
Study procedures:

* Consented at the time of enrollment in the study, which will be at hospital admission for delivery.
* Demographic data, medical history, obstetrical history, prenatal history and delivery information will be obtained from medical records and the subject
* Proteinuria, Placental weight, BMI, Birth weight and gender, mother smoker or not, clinical parameter of preeclampsia, and severity of preeclampsia, uterine artery Doppler results will be collected from medical records .
* SDF and NIRS application will be done once.

Measurements:

Sidestream dark field (SDF)

The side-stream darkfield camera ( CytoCam) will be put under the subjects tongue for 5-10 minutes. Multiple pictures of the small blood vessels will be taken.

Two fields will be selected that included at least 2 arterioles and 2 venules. Arterioles will be identified as high-flow vessels in which the direction of flow is from larger diameter vessels to smaller diameter vessels, while the reverse will be true for venules. Furthermore, arterioles will be distinguished from venules by the difference in erythrocyte flow velocity, which is substantially higher in arterioles than in venules. At least 2 arterioles and 2 venules will be taken from each captured image sequence to measure the blood vessel diameter.

The diameter of blood vessels will be determined using image processing software specifically designed for analysis of the microcirculation. The diameter of microvessels will be determined by drawing a perpendicular line from one side of the luminal vessel wall to the other at 3 separate locations. The functional capillary index (FCD) and the microvascular flow index (MFI) will be calculated as well. The FCD is defined as the total length of perfused capillaries per mm2. The MFI is used to describe the different flow velocities in venules in each observation field. This is a reproducible and validated index based on a semi-quantitative scoring (0=no flow, 1=intermittent flow, 2=sludging flow, 3=continuous flow and 4=high flow) of flow patterns in large (>50 μm), medium (25-50 μm) and small (10-25 μm, including capillaries) venules. Intermittent flow is characterized by a discontinuous flow pattern of erythrocytes during systolic heart contraction, which halts (or even reverses) during the diastolic phase. In sludging flow, individual erythrocytes have different low continuous velocities and they can be easily distinguished from each other. Continuous flow is characterized by an uninterrupted, uniform laminar flow pattern of erythrocytes that still just can be distinguished from each other. With high flow, the velocity of erythrocytes has exceeded the capture rate of the camera and therefore individual erythrocytes cannot be traced anymore and appear as a black column of cells.

CytoCam product is registered by the FDA with number D186803 Class1 exempt. This product is intended to be used for visualization of micro-circulation in tissue in orifices of the human body which may be non-invasively accessed and cutaneous surfaces.

Near-infra-red spectroscopy (NIRS) Artinis PortaLite with OxySoft softwear Artinis systems has developed a customizable NIRS device that measures tissue oxygenation saturation (StO2) of both muscle and brain tissue. This device can be customized in terms of emitter wavelength (5 are available, all in the NIR range) and configuration (2 emitters each @ 30, 35, and 40 mm from the detector). Critically, unlike most other commercially available NIRS devices for clinical care, the Artinis device allows exportation of the actual absorbance waveforms @ 15 Hz sampling rate. Thus, the Artinis PortaLite with OxySoft softwear will be used for research only, not for clinical care. The NIRS probe will be applied to one of the patient's thenar muscle and over the patient forehead and tissue oxygenation (TOI) will be recorded for 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older females (10 with diagnosis of preeclampsia and 10 with normal pregnancy),
* planned to deliver at UVA

Exclusion Criteria:

patients with:

* diabetes,
* gestational diabetes,
* gestational hypertension,
* chronic hypertension,
* chorioamniotitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age 18 years and older females (10 with diagnosis of preeclampsia and 10 with normal pregnancy), planned to deliver at UVA
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of microcirculatory changes by sidestream darkfield microscopy (SDF) | Day 1
  To assess whether sidestream darkfield microscopy (SDF) and could detect microcirculatory changes in patients who developed preeclampsia versus those who do not.
Tissue oxygenation assessed using Near-infra-red spectroscopy (NIRS) | Day 1
  Near-infra-red spectroscopy (NIRS),

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tiouririne, MD, Principal Investigator — University of Virginia Department of Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naljayan MV, Karumanchi SA. New developments in the pathogenesis of preeclampsia. Adv Chronic Kidney Dis. 2013 May;20(3):265-70. doi: 10.1053/j.ackd.2013.02.003. PMID 23928392
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Khan F, Belch JJ, MacLeod M, Mires G. Changes in endothelial function precede the clinical disease in women in whom preeclampsia develops. Hypertension. 2005 Nov;46(5):1123-8. doi: 10.1161/01.HYP.0000186328.90667.95. Epub 2005 Oct 17. PMID 16230524
- [Background] Anim-Nyame N, Gamble J, Sooranna SR, Johnson MR, Sullivan MH, Steer PJ. Evidence of impaired microvascular function in pre-eclampsia: a non-invasive study. Clin Sci (Lond). 2003 Apr;104(4):405-12. PMID 12653685
- [Background] Nama V, Manyonda IT, Onwude J, Antonios TF. Structural capillary rarefaction and the onset of preeclampsia. Obstet Gynecol. 2012 May;119(5):967-74. doi: 10.1097/AOG.0b013e31824ea092. PMID 22525907
- [Background] Pennings FA, Ince C, Bouma GJ. Continuous real-time visualization of the human cerebral microcirculation during arteriovenous malformation surgery using orthogonal polarization spectral imaging. Neurosurgery. 2006 Jul;59(1):167-71; discussion 167-71. doi: 10.1227/01.NEU.0000219242.92669.3B. PMID 16823313
- [Background] Mathura KR, Bouma GJ, Ince C. Abnormal microcirculation in brain tumours during surgery. Lancet. 2001 Nov 17;358(9294):1698-9. doi: 10.1016/S0140-6736(01)06722-8. PMID 11728549
- [Background] Perez-Barcena J, Goedhart P, Ibanez J, Brell M, Garcia R, Llinas P, Jimenez C, Ince C. Direct observation of human microcirculation during decompressive craniectomy after stroke. Crit Care Med. 2011 May;39(5):1126-9. doi: 10.1097/CCM.0b013e31820ead5e. PMID 21317640
- [Background] Sitina M, Turek Z, Parizkova R, Cerny V. In situ assessment of the brain microcirculation in mechanically-ventilated rabbits using sidestream dark-field (SDF) imaging. Physiol Res. 2011;60(1):75-81. doi: 10.33549/physiolres.931937. Epub 2010 Oct 15. PMID 20945959
- [Background] Diedler J, Zweifel C, Budohoski KP, Kasprowicz M, Sorrentino E, Haubrich C, Brady KM, Czosnyka M, Pickard JD, Smielewski P. The limitations of near-infrared spectroscopy to assess cerebrovascular reactivity: the role of slow frequency oscillations. Anesth Analg. 2011 Oct;113(4):849-57. doi: 10.1213/ANE.0b013e3182285dc0. Epub 2011 Aug 4. PMID 21821514
- [Background] Yamazaki K, Suzuki K, Itoh H, Muramatsu K, Nagahashi K, Tamura N, Uchida T, Sugihara K, Maeda H, Kanayama N. Cerebral oxygen saturation evaluated by near-infrared time-resolved spectroscopy (TRS) in pregnant women during caesarean section - a promising new method of maternal monitoring. Clin Physiol Funct Imaging. 2013 Mar;33(2):109-16. doi: 10.1111/cpf.12001. Epub 2012 Sep 23. PMID 23383688